CLINICAL TRIAL: NCT06813534
Title: " Contrast-free " IVUS Guided PCI Compared to Standard Angio-guided PCI in Patient With sEvere kidnEy Disease
Brief Title: IVUS Guided PCI in Patients With Chronic Kidney Disease
Acronym: SPEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230196
Record Dates: First submitted 2023-05-09; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; chronic kidney disease; Contrast induced nephropathy; IVUS
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventionnal PCI (Active Comparator): Contrast guided PCI
  Interventions: Device: Intravascular Ultrasound guided PCI
- IVUS guided PCI (Experimental): IVUS guided PCI with iodine contrast injection limited (as much as possible) to a final control injection.
  Interventions: Device: Intravascular Ultrasound guided PCI

INTERVENTIONS:
Device: Intravascular Ultrasound guided PCI — Intra-coronary ultrasound

SUMMARY:
The incidence of contrast-induced nephropathy (CIN) is high (> 25%) in patients with severe chronic renal disease (CKD) who undergo a percutaneous coronary procedure.

The development of CIN is a factor of poor prognosis and is associated with the occurrence of irreversible CKD, the need for dialysis, increased length of stay and hospital costs as well as the risk of death. There is no specific treatment for N-PCI, so its prevention is essential. Although many studies have been conducted to identify, compare and implement different pharmacological strategies for the prevention of CIN before percutaneous coronary procedurse, few per-procedural strategies have been studied to prevent this risk.

Intracoronary ultrasound (IVUS) is an essential tool, used routinely to guide percutaneous coronary procedures thanks to ultrasound, it does not require the injection of iodine contrast.

The main objective is to show that an IVUS-guided "zero-contrast" coronary angioplasty strategy in patients with severe renal impairment decreases the incidence of CIN within 72 hours of procedure.

DETAILED DESCRIPTION:
The incidence of contrast-induced nephropathy (CIN) is high (> 25%) in patients with severe chronic renal disease (CKD) who undergo a percutaneous coronary procedure.

The development of CIN is a factor of poor prognosis and is associated with the occurrence of irreversible CKD, the need for dialysis, increased length of stay and hospital costs as well as the risk of death. There is no specific treatment for N-PCI, so its prevention is essential. Although many studies have been conducted to identify, compare and implement different pharmacological strategies for the prevention of CIN before percutaneous coronary procedurse, few per-procedural strategies have been studied to prevent this risk.

Intracoronary ultrasound (IVUS) is an essential tool, used routinely to guide percutaneous coronary procedures thanks to ultrasound, it does not require the injection of iodine contrast.

The main objective is to show that an IVUS-guided "zero-contrast" coronary angioplasty strategy in patients with severe renal impairment decreases the incidence of CIN within 72 hours of procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Indication for PCI
* Chronic kidney disease with creatinine clearance ≤ 30 mL/min/1.73m²
* Feasibility of IVUS determined by 2 trained interventional cardiologist
* Affiliated to social security

Exclusion Criteria:

* Iodine contrast injection in the previous 72 hours
* Known allergy to iodine contrast
* Permanent dialysis
* Chronic total occlusion
* Hemodynamic instability
* Legal protection
* Pregnant of breastfeeding patients
* Patients on "AME"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2027-07-07 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
Rate of serum creatinine due to nephropathy | 30 days
  Contrast-induced nephropathy is defined as an increase in creatininemia by 25% from its baseline level. The parameter being measured is creatininemia, which refers to the concentration of creatinine in the blood. The unit of measurement for this increase is a percentage (%)

SECONDARY OUTCOMES:
Global safety | 30 days
  The occurrence of death from any cause within 30 days. The unit of measurement is the presence or absence of death.
Endocoronary complications | 72 hours
  his includes dissection, thrombus formation, breaches, or coronary occlusion that require an additional unplanned intervention. The unit of measurement is the occurrence of these complications, recorded as Yes or No.
Procedural Criteria | 72 hours
  Procedure time: The total time taken for the procedure. The unit of measurement is time, typically recorded in minutes (min)
Myocardial infarction | 30 days
  The occurrence of a myocardial infarction within 30 days. The unit of measurement is the presence or absence of the event, recorded as Yes or No."
Global safety : stroke | 30 days
  Stroke: The occurrence of a stroke within 30 days. The unit of measurement is the presence or absence of the event, recorded as Yes or No
Global safety | 30 days
  Unplanned hospitalization for cardiac or renal causes: The occurrence of an unplanned hospitalization due to cardiac or renal causes within 30 days. The unit of measurement is the presence or absence of the event, recorded as Yes or No.
Angioplasty failures | 72 hours
  Angioplasty failures are defined by a residual stenosis of 70% or greater and/or a TIMI flow of less than 3 at the end of the procedure. The unit of measurement for residual stenosis is percentage (%) and for TIMI flow, the unit is a scale from 0 to 3, with a TIMI flow of less than 3 indicating failure.
Procedural Criteria : Fluoroscopy time | 72 hours
  Fluoroscopy time: The amount of time fluoroscopy imaging is used during the procedure. The unit of measurement is time, typically recorded in minutes (min)
Procedural Criteria: Air Kerma | 72 hours
  Air Kerma: A measure of the radiation dose delivered during the procedure. The unit of measurement is the Gray (Gy), specifically milligray (mGy) for this context
Procedural Criteria : PDS (Procedure Dose Score) | 72 hours
  PDS (Procedure Dose Score): A measure of the total radiation dose delivered to the patient during the procedure. The unit of measurement is arbitrary units based on the specific scoring system used.
Procedural Criteria | 72 hours
  Volume of contrast injected: The amount of contrast material used during the procedure. The unit of measurement is milliliters (mL)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Romain GALLET, Créteil, Creteil
  - Romain GALLET, Créteil

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION